CLINICAL TRIAL: NCT05102552
Title: A Single-Center, Randomized, Open-label, Multiple-Dose, Single-Sequence Crossover Study, Evaluating the Safety and Relative Bioavailability of Three SPN-817 Treatments (A, B and C) in Healthy Adult Subjects
Brief Title: Evaluating the Safety and Relative Bioavailability of Three SPN-817 Treatments (A, B and C) in Healthy Adult Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 817P106
Record Dates: First submitted 2021-09-22; First posted 2021-11-01 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — huperzine A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): BIS-001: Treatment A and SPN-817: Treatment B
  Interventions: Drug: SPN-817, Treatment B; Drug: BIS-001, Treatment A
- Cohort 2 (Active Comparator): BIS-001: Treatment A and SPN-817: Treatment C
  Interventions: Drug: SPN-817, Treatment C; Drug: BIS-001, Treatment A

INTERVENTIONS:
Drug: SPN-817, Treatment B — SPN-817 Treatment B, is an Extended Release formulation of Huperzine A, an acetylcholinesterase inhibitor
  Other Names: Huperzine A
  Arms: Cohort 1
Drug: SPN-817, Treatment C — SPN-817 Treatment C, is an Extended Release formulation of Huperzine A, an acetylcholinesterase inhibitor
  Other Names: Huperzine A
  Arms: Cohort 2
Drug: BIS-001, Treatment A — BIS-001 is an Extended Release formulation of Huperzine A, an acetylcholinesterase inhibitor
  Other Names: Huperzine A

SUMMARY:
Randomized, Open-Label, Multiple Dose study to evaluate the relative bioavailability of Treatment A, Treatment B, and Treatment C

DETAILED DESCRIPTION:
A Single-Center, Randomized, Open-label, Multiple-Dose, Single-Sequence Crossover Study, Evaluating the Safety and Relative Bioavailability of Three SPN-817 Treatments (A, B and C) in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria

1. Healthy adult male or female volunteers, 18-55 years of age inclusive.
2. Weight of at least 50 kg and within the normal Body Mass Index (BMI) between 18 - 32 kg/m2 (inclusive).
3. Considered medically healthy by the Investigator via assessment of physical and neurological examinations, medical history, clinical laboratory tests, vital signs, and electrocardiogram (ECG)
4. Able and willing to swallow whole capsules and capsule contents without breaking, cutting, or chewing.
5. Able to voluntarily provide written informed consent to participate in the study.
6. Post-menopausal females with amenorrhea for at least 12 months with a serum follicle stimulating hormone [FSH] level of >40 IU/L) or women of non-childbearing potential (WONCBP) who are permanently sterilized (bilateral tubal ligation, hysterectomy, bilateral oophorectomy for six months minimum prior to screening).
7. Non-pregnant females of childbearing potential who are either sexually inactive (abstinent) or, if sexually active with a male partner who is biologically capable of having children, agree to use one of the following acceptable birth control methods beginning 14 days prior to the first dose, throughout the study, and for 30 days following the last dose:

   * Hormonal contraceptive (i.e., oral, transdermal/subdermal; implant or injection)
   * Intrauterine device (IUD)
   * Double contraceptive methods (e.g. oral contraception and condom)
   * Vasectomized partner (6 months minimum)
8. Male subjects who are biologically capable of having children (i.e., non-vasectomized) who are sexually inactive (abstinent) or, if sexually active with a female of childbearing potential, must agree to use one or more of the above forms of birth control for themselves and their partner(s), as appropriate, beginning 14 days prior to the first dose through at least 90 days following the last administration of study drug. They must also agree to abstain from sperm donation from the first administration of study drug to 90 days after the last administration of study drug.

Exclusion Criteria

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
2. Evidence of suicidality (defined as either active suicidal plan/intent or active suicidal thoughts, or more than one lifetime suicide attempt) within six months before Screening, or at Screening and Day -1 as determined by C-SSRS.
3. Evidence of infection with Hepatitis B or C, or human immunodeficiency virus HIV-1 or HIV2, as determined by results of testing at screening.
4. Positive urine drug screen (for amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, tetrahydrocannabinol and phencyclidine) at Screening and at Day -1.
5. Clinically significant cardiology abnormalities at Screening and Day -1.

   * Abnormal ECG that is, in the investigator's opinion, clinically significant including heart rate <50 BPM (average of 3);
   * PR interval > 220 ms;
   * QRS interval ≥ 120 ms;
   * QTcF interval > 450 ms (QT corrected using Fridericia's method);
   * Second or third-degree atrioventricular block;
   * Any rhythm, other than sinus rhythm, that is interpreted by the investigator to be clinically significant.
6. Creatinine clearance < 80 mL/min, according to the Cockcroft-Gault equation at Screening or Day -1.
7. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate [HR] less than 50 or over 100 bpm) at Screening or check-in on Day -1.
8. History of intellectual disability (intellectual developmental disorder) or mental retardation.
9. A history of neuroleptic malignant syndrome.
10. A history of cancer within 5 years prior to screening or between screening and randomization (with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin), any history of renal cell carcinoma or breast cancer, or a family history of lymphangioleiomyomatosis in association with tuberous sclerosis complex (TSC-LAM).
11. A history of clinically significant head trauma, including closed head injury with loss of consciousness.
12. A history of seizure, loss of consciousness for an unknown reason, or any other known neurological disorder placing the subject at risk for seizures.
13. History of significant alcohol abuse or drug abuse within one year prior to screening.
14. Regular use of alcohol within six months prior to Screening (more than 14 units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test at Screening or Day -1.
15. Use of drugs of abuse (such as cocaine, phencyclidine, amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, tetrahydrocannabinol and phencyclidine ) within one year prior to Screening, or positive urine drug screen (for amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, tetrahydrocannabinol and phencyclidine) at Screening or Day -1.
16. History of an allergic reaction to investigational product or related drugs, such as those with similar mechanism of action.
17. History of previous exposure to investigational product in a clinical trial.
18. Female subjects who are pregnant or lactating.
19. Use of prescription medication within 14 days prior to administration of study drug, or over-the-counter products (including natural food supplements) within seven days prior to administration of study drug. Exceptions include topical products without systemic absorption, hormonal contraceptives, hormone replacement therapy (stable dose for at least 30 days), and acetaminophen (2 g/day).
20. Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
21. History of anaphylaxis or severe allergy to any drug, food, toxin, or other exposure.
22. Subjects who received any investigational drug, device or biologic within 3 months or 5 half-lives (whichever is longer) of Day 1 dosing of study drug.
23. Subjects who have had the following blood or plasma donation:

    * Subjects who donated 50 to 499mL of blood within 30 days and more than 499mL within 56 days prior to the first dose or have hemoglobin <128 g/L (males) or <115 g/L (females) and hematocrit <0.37 L/L (males) or <0.32 L/L (females) at Screening.
    * Subjects who have had donated plasma within 7 days prior to dosing
24. Tobacco use as indicated by > 5 cigarettes per week or the equivalent, 30 days prior to Day -1.
25. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability | 22 days
  Area under the curve (AUC)
Relative Bioavailability | 22 days
  Peak (Cmax) plasma concentration

SECONDARY OUTCOMES:
To assess the safety and tolerability of multiple oral administration of SPN-817 in healthy adult subjects. | 25 days
  Adverse Events (occurrence/incidence, seriousness, severity, and causality assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanelle Portelli, Ph.D., Study Director — Supernus Pharmaceuticals
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No